CLINICAL TRIAL: NCT05881538
Title: Effectiveness of a High-intensity Intervallic Training Program in Children and Adolescents With Post-infectious Bronchiolitis Obliterans: a Randomized Controlled Trial
Brief Title: High Intensity Intervallic Training in Children With Bronchiolitis Obliterans
Acronym: PIBOHIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Consejo Superior de Deportes, Spain (Other)
Responsible Party: Principal Investigator, Márcio Vinícius Fagundes Donadio, Professor, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PIBOHIIT-UIC
Record Dates: First submitted 2023-04-24; First posted 2023-05-31 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Bronchiolitis Obliterans
Keywords: High intensity interval training; Post-infectious bronchiolitis obliterans; Telematic program; Cardiorespiratory fitness
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Multicenter study, randomized controlled trial in two parallel groups (ratio 1:1), double blinded.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The evaluators and care providers will be masked to the allocation of the patients. Given the nature of the intervention, it is not possible to mask patients or monitors in charge of supervising the execution of the exercise training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): 16 weeks of a "High Intensity Interval Training" exercise program conducted telematically with real time supervision twice a week.
  The exercise program consists of a circuit of exercises aiming to achieve a target heart rate for each fitness level.
  Interventions: Other: Exercise group
- Control group (No Intervention): Routine physician recommendations for physical activity.

INTERVENTIONS:
Other: Exercise group — Participants will perform a 16-week High Intensity Interval Training exercise program, twice a week. The intervention will be conducted telematically with real time supervision.
  Other Names: High Intensity Interval Training
  Arms: Exercise group

SUMMARY:
Post-Infectious Bronchiolitis Obliterans (PIBO) is an irreversible obstructive lung disease characterized by subepithelial inflammation and fibrotic narrowing of the bronchioles after lower respiratory tract infection. This disease is diagnosed mainly in children, more frequently before the age of 2 years. Due to symptoms such as dry cough and dyspnea sensation, most of these patients have low levels of physical activity compared to healthy individuals. Physical activity can positively influence oxygen consumption, muscle strength, and quality of life. High levels of oxygen consumption are associated with a lower risk of respiratory disease and hospitalization. High-intensity interval training (HIIT) may be an effective way to improve oxygen consumption, muscle strength, and quality of life in patients with chronic diseases. HIIT has been shown to produce less dyspnea sensation and to be more entertaining in children and adolescents with respiratory disease compared to continuous training. Thus, the investigators propose to perform telematically real-time guided training to reduce travel times and additional costs to patients.

Objective: To analyze the effects of a telematically supervised high-intensity intervallic training program on aerobic fitness, as well as functional/clinical outcomes in patients with PIBO.

Methods: Randomized controlled trial with two groups. Exercise group: 16-week HIIT training conducted telematically; Control group: will follow the routine physician's recommendations. Patients will be recruited at Vall D'Hebrón University Hospital (Barcelona), Niño Jesús University Hospital (Madrid), and Donostia Universitary Hospital (San Sebastián). Criteria for participation: (I) Diagnosis of PIBO; (II) Clinically stable at the time of the assessments; (III) Age between 6 to 20 years old.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Postinfectious bronchiolitis obliterans;
* Clinical stability at the time of the assessments;
* Age between 6 and 20 years old.

Exclusion Criteria:

* Symptoms of pulmonary exacerbation during the last four weeks;
* Diagnosis of other cardiorespiratory diseases leading to symptoms of persistent respiratory dysfunction;
* Difficulty in comprehension or musculoskeletal alterations that may influence the assessments;
* Pregnancy;
* Transplant list inclusion.

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen consumption | Change from baseline to 16 weeks
  Change in peak oxygen consumption (mL/kg/min) will be evaluated through cardiopulmonary exercise testing (CPET).
Change in time to ventilatory threshold | Change from baseline to 16 weeks
  Change in time to ventilatory threshold (minutes) will be evaluated through cardiopulmonary exercise testing (CPET).
Change in percent oxygen consumption at ventilatory threshold | Change from baseline to 16 weeks
  Change in percent oxygen consumption at ventilatory threshold will be evaluated through cardiopulmonary exercise testing (CPET).
Change in ventilatory efficiency | Change from baseline to 16 weeks
  Change in ventilatory efficiency will be evaluated by combining ventilation (VE) and carbon dioxide production (VCO2) measurements to report VE/VCO2 ratio, evaluated through cardiopulmonary exercise testing (CPET).

SECONDARY OUTCOMES:
Change in forced expiratory volume in the first second | Change from baseline to 16 weeks
  Change in forced expiratory volume in the first second (liters) will be evaluated through spirometry.
Change in forced vital capacity | Change from baseline to 16 weeks
  Change in forced vital capacity (liters) will be evaluated through spirometry.
Change in forced expiratory flow between 25 and 75% of forced vital capacity | Change from baseline to 16 weeks
  Change in forced expiratory flow between 25 and 75% of forced vital capacity (liters/minute) will be evaluated through spirometry.
Change in muscle strength | Change from baseline to 16 weeks
  Changes in muscle strength will be evaluated using a dynamometer.
Change in lower body strength | Change from baseline to 16 weeks
  Changes in lower body strength will be evaluated using the 30 seconds Sit to Stand Test (30STS).
Change in free fat mass | Change from baseline to 16 weeks
  Changes in free fat mass (percent) will be evaluated through bioimpedance.
Change in lean mass | Change from baseline to 16 weeks
  Changes in lean mass (percent) will be evaluated through bioimpedance.
Change in hip-waist ratio | Change from baseline to 16 weeks
  Changes in hip-waist ratio will be evaluated by combining hip circumference and waist circumference measurements using a non-stretchable tape measure.
Change in body mass index | Change from baseline to 16 weeks
  Changes in body mass index will be evaluated by combining weight and height measurements to report BMI (kg/m^2).
Change in quality of life | Change from baseline to 16 weeks
  Changes in quality of life will be evaluated through the Saint George's Respiratory Questionnaire (SRQ). The overall result of the scale is a numerical value from 0 to 100, with the highest values corresponding to a worse quality of life.
Change in dyspnea | Change from baseline to 16 weeks
  Changes in dyspnea will be evaluated through the Medical Research Council (mMRC) modified dyspnea scale. The overall result of the scale is a numerical value from 0 to 4, where the highest value corresponds to the worse dyspnea.

OTHER OUTCOMES:
Height in meters | Change from baseline to 16 weeks
  Height will be evaluated using a stadiometer.
Weight in kilograms | Change from baseline to 16 weeks
  Weight will be evaluated using a weight scale.
Daily physical activity level | Change from baseline to 16 weeks
  Daily physical activity level will be evaluated through the physical activity questionnaire (PAQ). The overall test score is from 1 to 5 points, with a higher score indicating a higher level of activity.

CONTACTS AND LOCATIONS:
Overall Officials: Márcio VF Donadio, PhD, Principal Investigator — Universitat Internacional de Catalunya
Locations (3):
- Spain (3):
  - Hospital Universitario Donostia, Donostia / San Sebastian, Basque Country
  - Hospital Universitari Vall d'Hebron, Barcelona, Catalonia
  - Hospital Universitario Infantil Niño Jesús, Madrid

IPD SHARING:
Plan to Share IPD: Yes
The investigators will collect patients' personal data and clinical history by means of the information delivered by the participating hospital. These data will be stored and coded in an Excel file in order to protect confidentiality before, during and after the study. All information will be entered and stored electronically in the institutional platform REDCAP hosted on the hospitals' server.
Time Frame: After completion of study, the data will be stored for as long as necessary to meet any possible responsibilities derived from the study.
Access Criteria: Access will be given only to the researchers of the study.

DOCUMENTS (1):
  • Informed Consent Form (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT05881538/ICF_000.pdf